CLINICAL TRIAL: NCT02523183
Title: The Use of Medicinal Cannabinoids as Adjunctive Treatment for Medically Refractory Epilepsy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Colorado, Denver (Other)
Collaborators: Colorado Department of Public Health and Environment (Other Government)
Responsible Party: Sponsor
Other Study IDs: 14-1606
Record Dates: First submitted 2015-07-23; First posted 2015-08-14 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Epilepsy, Unspecified, Refractory (Medically)
Keywords: Epilepsy; Marijuana
MeSH Terms: conditions — Epilepsy; Marijuana Abuse | interventions — Medical Marijuana

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples will be collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects with medically refractory epilepsy: Pediatric epilepsy patients who are followed at Children's Hospital Colorado with medically refractory epilepsy, and whom the family has decided to treat with medical cannabis.
  Interventions: Drug: Medical Cannabis

INTERVENTIONS:
Drug: Medical Cannabis — Pediatric patients with medically refractory epilepsy and treated with medicinal cannabis.
  Other Names: medicinal cannabinoids (MCBD)

SUMMARY:
Many families of children with medically refractory epilepsy are choosing to use medicinal cannabinoids (MCBD) as an adjunctive alternative treatment option. The safety, tolerability and efficacy of these products are not known. The primary objective of this study is to determine how the use of MCBD affects children with medically refractory epilepsy in an observational study. Measures of evaluation to be used will include: laboratory values, developmental measures, seizure diaries and serial electroencephalographic (EEG) recordings.

DETAILED DESCRIPTION:
This is an observational study of a family's choice to use MCBD and the effect of this substance on medically refractory epilepsy in children. The risks associated with this use are not well known. There have recently been reports of stroke, liver dysfunction and altered anticonvulsant levels. In addition, there have been long term risks reported of decreased memory function, cognitive problems and executive function abnormalities. This study does not condone or advocate the use of the substance but merely seeks to document the short term effects of the use in this population. It should be noted that providers at Children's Hospital Colorado are not registered providers for medicinal cannabis; therefore, this will be an observational study of effects of this substance as prescribed by other physicians outside of our institution.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female >1 month of age
2. Documentation of a diagnosis of medically refractory epilepsy as evidenced by medical records, genetic testing and/or the following clinical features:

   * Failure to control seizures despite an appropriate trial of two anticonvulsant medications at therapeutic doses
3. Baseline seizure frequency of at least 2 per week of the any of the following types:

   * Generalized tonic-clonic
   * Clonic
   * Tonic
   * Hemiconvulsive
   * Drop attacks
   * Focal motor
   * Epileptic spasms
4. 1-3 baseline anti-seizure medications at stable doses for a minimum of 4 weeks prior to enrollment.
5. Written informed consent obtained from the patient or the patient's legal representative.

Exclusion Criteria:

1. Epilepsies associated with rapidly progressing neurodegenerative diseases ex: Rasmussen encephalitis, and tumors.
2. Epilepsies associated with treatable inborn errors of metabolism
3. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
4. Non-epileptic events.
5. Current use of MCBD products (Note: Patient is eligible if currently using MCBD but will be switching to a different product).

Ages: 1 Month to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric epilepsy patients who are followed at Children's Hospital Colorado with medically refractory epilepsy, and whom the family has decided to treat with medicinal cannabis. Children who have not been treated with medically accepted standard treatment for their epilepsy condition will not be accepted into this study as the researchers do not want to be misperceived as condoning the use of medical marijuana in lieu of standard treatment.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2015-07; Primary Completion 2020-10 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in background and architecture of seizures confirmed by non-investigational EEG | Baseline, 4 weeks, 8 weeks, and 12 weeks
  Prolonged EEG recordings lasting 24-48 hours (whichever is clinically indicated) will be performed in either the home setting as an ambulatory EEG or in the hospital in the Epilepsy Monitoring Unit. This decision will be made on a clinical basis. This will allow for objective quantification of seizures in children with frequent seizures that occur on a daily basis and background EEG changes for other children. Two EEGs will be done: one at baseline, and one at the end of the study.
Seizure Frequency | Baseline, 4 weeks, 8 weeks, and 12 weeks
  Each subject will maintain a seizure diary. Rescue drug use and VNS (Vagus Nerve Stimulation) activations will be tracked as an adjunct to all current anti-seizure medications. Frequency of status epilepticus will be tracked as well as hospital visits for seizures or adverse events from MCBD. Clinical evaluations will be taken every 2 months throughout the duration of the study. Subjects will be monitored every 2 weeks by telephone and/or email.
Pediatric Epilepsy Side Effects Questionnaire | Baseline, 4 weeks, 8 weeks, and 12 weeks
  Side effects will be evaluated using PESQ (Pediatric epilepsy Side Effects Questionnaire). This questionnaire will be administered 4 weeks, 8 weeks, and 12 weeks after baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Knupp, MD, Principal Investigator — Assistant Professor of Pediatrics and Neurology
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

REFERENCES:
- See also: More information about medical marijuana research at childrens hospital colorado — http://www.childrenscolorado.org/wellness-safety/parent-resources/marijuana-what-parents-need-to-know/research